CLINICAL TRIAL: NCT05294445
Title: From the Emergency Department Directly to Ablation of Atrial Fibrillation - Study - The "EMERGE-Cryo-Study"
Brief Title: From the Emergency Department Directly to Ablation of Atrial Fibrillation Study
Acronym: EMERGE-Cryo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asklepios proresearch (Industry)
Collaborators: Atrial Fibrillation Network (Other); Medtronic Bakken Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #3794
Record Dates: First submitted 2022-03-04; First posted 2022-03-24 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: prospective, two-arm, randomized, open-label, blinded endpoint, multi-center study
Who Masked: Outcomes Assessor
Masking Description: Additionally to ILR interrogation on each site, the ILR data will be reviewed by blinded core lab investigators. All observed primary endpoints and outcome parameters will be presented to ERC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group1: Cryo-AF-Ablation (Active Comparator): Patients randomized in the Cryo-AF-Ablation group should receive the cryo AF ablation within 21 days from baseline.
  Interventions: Procedure: Ablation of atrial fibrillation (AF)
- Group 2: Usual care (No Intervention): Patients randomized in the usual care group should start or maintain on AAD therapy within 21 days from baseline, based on decision of the investigator according to current ESC Guidelines.

INTERVENTIONS:
Procedure: Ablation of atrial fibrillation (AF) — Cryo-AF-ablation of pulmonary vein (pulmonary vein isolation = PVI)
  Arms: Group1: Cryo-AF-Ablation

SUMMARY:
The study is a prospective, two-arm, randomized, open-label, blinded endpoint, multi-center study to investigate the impact of first line ablation in patients presenting at the emergency room with recent-onset paroxysmal or persistent atrial fibrillation.

DETAILED DESCRIPTION:
As stated in the current guidelines, the prevalence of AF tripled over the last 30 years and further progress is expected. AF is associated with increased mortality and morbidity. Approximately 70% of the patients who are hospitalized for AF are admitted through the emergency department. The steady increase of AF-related visits at the emergency departments therefore lead to a high number of hospitalizations. The direct costs of AF already amount to approximately 1% of total healthcare spending, driven by AF-related complications (e.g. stroke) and treatment costs (e.g. hospitalizations). These costs will increase dramatically unless AF is prevented and treated in a timely and effective manner.

Catheter ablation therapy has been proven to be safe and effective for the treatment of paroxysmal and persistent AF and is now standard in AF therapy. Several trials have shown that catheter ablation of AF is superior to antiarrhythmic drug therapy. As evidenced by the FIRE & ICE trial, cryoballoon ablation is non-inferior to the former goldstandard of radiofrequency current (RFC) energy. Importantly, it has been reported that cryoballoon ablation was associated with a reduction in resource use and costs as compared to RFC ablation of AF. These cost savings persisted over multiple healthcare systems.

However, data on the optimal timing of AF ablation is scarce. While there is evidence that catheter ablation is highly efficient in delaying progression from paroxysmal to persistent AF, there are only few trials evaluating a strategy of early treatment of AF, regarding the patients' medical history (CRYO-FIRST, EARLY-AF). Another trial investigated the utilization of a multidisciplinary AF treatment pathway in patients presenting to the emergency department, which resulted in reduction of admission rate and hospital stays but did not include catheter ablation of AF. However, there is no scientific evidence on a strategy of early treatment of atrial fibrillation comparing anti-arrhythmic drug therapy to catheter ablation in the large number of patients presenting to the emergency departments.

A well-known limitation of many trials investigating catheter ablation of AF, can be found during the trials follow up after ablation, as detection of AF recurrences can be challenging. The sensitivity of detecting asymptomatic episodes with intermittent 24-hours ECG-monitoring is low. The Heart Rhythm Society and the European Heart Rhythm Society encourage continuous arrhythmia monitoring due to the greater sensitivity in detecting symptomatic and asymptomatic AF recurrences but also when assessing the overall AF burden. Additionally, in an era of digital revolution, the AFNET incorporated the use of wearables, smartphones, hand held-devices and health-related apps to new approaches of AF management.

To evaluate the efficacy and safety of an early rhythm control treatment of AF by catheter ablation with the cryoballoon with particular respect to arrhythmia recurrence, rehospitalisation, heart failure and health care costs in patients presenting to the emergency department due to AF, a prospective randomized study is necessary.

ELIGIBILITY:
Inclusion Criteria:

* Documented, paroxysmal or persistent AF (longest AF episode < 6-month duration). Any ECG documentation of AF (12 lead ECG, Holter ECG or mobile ECG monitoring) needs to be presented.
* Recent-onset AF (≤ 1 year prior to enrolment)
* Presenting at the emergency department or outpatient clinic within the last 2 weeks because of AF, including patients with spontaneous conversion in sinus rhythm (with prior AF documentation)
* Age ≥ 18 years
* Subject is able and willing to give informed consent

Exclusion Criteria

* Pers. AF > 6 Mon (one episode)
* LA-Diameter > 60mm
* Severe mitral stenosis or regurgitation, prior mitral valve reconstruction or replacement
* Any previous left atrial ablation
* Ongoing continuous AAD therapy with Amiodarone at baseline
* History of failed continuous AAD therapy with > 1 agent. Exceptions are Beta blocker, Verapamil or "pill in the pocket"-therapy.
* Any condition or disease, which is contraindication for AF ablation, up to the assessment of the investigator
* Any condition or disease, which is a contraindication for antiarrhythmic drug treatment, up to the assessment of the investigator
* Known intra-cardiac thrombus formation under continuous oral anticoagulation (defined as intake >4 weeks)
* Any contraindication for oral anticoagulation
* Any untreated or uncontrolled hyperthyroidism or other reversible causes for AF like alcoholism
* Pregnant or breastfeeding woman or woman of childbearing potential not on adequate birth control
* Active systemic infection
* Co-Existence of non PV-dependent atrial Tachycardia
* Indication for implantation of ICD or pacemaker

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-12-14 (Estimated); Study Completion 2028-12-14 (Estimated)

PRIMARY OUTCOMES:
Freedom from any atrial tachyarrhythmia | within 3 to 12 months follow-up
  Freedom from any atrial tachyarrhythmia, including atrial fibrillation (AF), atrial flutter and atrial tachycardias (>30 s) through 3 to 12 months follow-up on ILR monitoring or any 12 lead ECG on visits, ECG Holter monitoring, or on symptom driven event monitoring

SECONDARY OUTCOMES:
AF burden (1) | within 3 to 12 months follow up
  AF burden between 3 to 12 months after randomization. AF burden is defined as overall percentage of AF during the observed time
AF burden (2) | within 0 to 12 months follow up
  AF burden between 0 to 3, 3 to 6 and 6 to 12 months after randomization
Freedom from atrial fibrillation | within 3 to 12 months follow up
  Freedom from atrial fibrillation (AF) (>30 s)
Freedom from atrial tachycardia and atrial flutter | within 3 to 12 months follow up
  Freedom from atrial tachycardia and atrial flutter (AFl)
symptomatic versus asymptomatic atrial tachyarrhythmia | within 3 to 12 months follow up
  Analysis of amount of symptomatic versus asymptomatic atrial tachyarrhythmia recurrences
Re-hospitalization rate | up to 12 months follow up
  Re-hospitalization rate due to cardiovascular disease (AF, worsening of heart failure, cardiovascular disease)
Progression of heart failure | up to 12 months follow up
  Progression of heart failure defined as trend in LV-EF and trend in BNP
Quality of life (AFEQT and EQ-5D-5L) | within 0 to 12 months follow up
  Improvement of quality of life at 12 months compared to baseline (AFEQT and EQ-5D-5L Questionnaire)
Safety / Complications | within 0 to 12 months follow up
  Safety / Complications

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Willems, MD, PhD, Principal Investigator — Asklepios Hospital St. Georg, Hamburg, Germany
Locations (13):
- Germany (13):
  - Asklepios Klinik St. Georg, Hamburg, Hamburg
  - Universitäres Herz- und Gefäßzentrum, Hamburg, Hamburg
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Deutsches Herzzentrum der Charité, Berlin
  - Herzzentrum Uniklinik Köln, Cologne
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - Cardioangiologisches Zentrum Bethanien (CCB) am Markuskrankenhaus, Frankfurt
  - Universitätsklinikum Giessen, Giessen
  - AK Altona, Hamburg
  - AK Nord, Hamburg-Nord
  - Asklepios Klinik Harburg, Harburg
  - Universitätsklinikum Münster, Münster
  - St. Josefs-Hospital Wiesbaden GmbH, Wiesbaden

REFERENCES:
- [Background] Packer DL, Mark DB, Robb RA, Monahan KH, Bahnson TD, Poole JE, Noseworthy PA, Rosenberg YD, Jeffries N, Mitchell LB, Flaker GC, Pokushalov E, Romanov A, Bunch TJ, Noelker G, Ardashev A, Revishvili A, Wilber DJ, Cappato R, Kuck KH, Hindricks G, Davies DW, Kowey PR, Naccarelli GV, Reiffel JA, Piccini JP, Silverstein AP, Al-Khalidi HR, Lee KL; CABANA Investigators. Effect of Catheter Ablation vs Antiarrhythmic Drug Therapy on Mortality, Stroke, Bleeding, and Cardiac Arrest Among Patients With Atrial Fibrillation: The CABANA Randomized Clinical Trial. JAMA. 2019 Apr 2;321(13):1261-1274. doi: 10.1001/jama.2019.0693. PMID 30874766
- [Background] Asad ZUA, Yousif A, Khan MS, Al-Khatib SM, Stavrakis S. Catheter Ablation Versus Medical Therapy for Atrial Fibrillation: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Circ Arrhythm Electrophysiol. 2019 Sep;12(9):e007414. doi: 10.1161/CIRCEP.119.007414. Epub 2019 Aug 21. PMID 31431051
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] Gunawardene MA, Hoffmann BA, Schaeffer B, Chung DU, Moser J, Akbulak RO, Jularic M, Eickholt C, Nuehrich J, Meyer C, Willems S. Influence of energy source on early atrial fibrillation recurrences: a comparison of cryoballoon vs. radiofrequency current energy ablation with the endpoint of unexcitability in pulmonary vein isolation. Europace. 2018 Jan 1;20(1):43-49. doi: 10.1093/europace/euw307. PMID 27742775
- [Background] Gunawardene MA, Hartmann J, Jularic M, Eickholt C, Gessler N, Willems S. [Therapeutic management of nonvalvular atrial fibrillation]. Herz. 2020 Sep;45(6):603-616. doi: 10.1007/s00059-020-04960-w. German. PMID 32632547
- [Background] Gunawardene MA, Eickholt C, Akbulak RO, Jularic M, Klatt N, Hartmann J, Schluter M, Meyer C, Willems S, Schaeffer B. Ultra-high-density mapping of conduction gaps and atrial tachycardias: Distinctive patterns following pulmonary vein isolation with cryoballoon or contact-force-guided radiofrequency current. J Cardiovasc Electrophysiol. 2020 May;31(5):1051-1061. doi: 10.1111/jce.14413. Epub 2020 Mar 9. PMID 32107811
- [Background] Schmidt M, Dorwarth U, Andresen D, Brachmann J, Kuck KH, Kuniss M, Lewalter T, Spitzer S, Willems S, Senges J, Junger C, Hoffmann E. Cryoballoon versus RF ablation in paroxysmal atrial fibrillation: results from the German Ablation Registry. J Cardiovasc Electrophysiol. 2014 Jan;25(1):1-7. doi: 10.1111/jce.12267. Epub 2013 Oct 17. PMID 24134539
- [Background] Dinshaw L, Schaffer B, Akbulak O, Jularic M, Hartmann J, Klatt N, Dickow J, Gunawardene M, Munkler P, Hakmi S, Pecha S, Sultan A, Luker J, Pinnschmidt H, Hoffmann B, Gosau N, Eickholt C, Willems S, Steven D, Meyer C. Long-term efficacy and safety of radiofrequency catheter ablation of atrial fibrillation in patients with cardiac implantable electronic devices and transvenous leads. J Cardiovasc Electrophysiol. 2019 May;30(5):679-687. doi: 10.1111/jce.13890. Epub 2019 Mar 10. PMID 30821012
- [Background] Stewart S, Murphy NF, Walker A, McGuire A, McMurray JJ. The current cost of angina pectoris to the National Health Service in the UK. Heart. 2003 Aug;89(8):848-53. doi: 10.1136/heart.89.8.848. PMID 12860855
- [Background] Jackson SL, Tong X, Yin X, George MG, Ritchey MD. Emergency Department, Hospital Inpatient, and Mortality Burden of Atrial Fibrillation in the United States, 2006 to 2014. Am J Cardiol. 2017 Dec 1;120(11):1966-1973. doi: 10.1016/j.amjcard.2017.08.017. Epub 2017 Aug 30. PMID 28964382
- [Background] Ptaszek LM, Baugh CW, Lubitz SA, Ruskin JN, Ha G, Forsch M, DeOliveira SA, Baig S, Heist EK, Wasfy JH, Brown DF, Biddinger PD, Raja AS, Scirica B, White BA, Mansour M. Impact of a Multidisciplinary Treatment Pathway for Atrial Fibrillation in the Emergency Department on Hospital Admissions and Length of Stay: Results of a Multi-Center Study. J Am Heart Assoc. 2019 Sep 17;8(18):e012656. doi: 10.1161/JAHA.119.012656. Epub 2019 Sep 12. PMID 31510841
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Heart Rhythm. 2017 Oct;14(10):e275-e444. doi: 10.1016/j.hrthm.2017.05.012. Epub 2017 May 12. No abstract available. PMID 28506916
- [Background] Hakalahti A, Biancari F, Nielsen JC, Raatikainen MJ. Radiofrequency ablation vs. antiarrhythmic drug therapy as first line treatment of symptomatic atrial fibrillation: systematic review and meta-analysis. Europace. 2015 Mar;17(3):370-8. doi: 10.1093/europace/euu376. Epub 2015 Feb 1. PMID 25643988
- [Background] Kuck KH, Brugada J, Furnkranz A, Metzner A, Ouyang F, Chun KR, Elvan A, Arentz T, Bestehorn K, Pocock SJ, Albenque JP, Tondo C; FIRE AND ICE Investigators. Cryoballoon or Radiofrequency Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2016 Jun 9;374(23):2235-45. doi: 10.1056/NEJMoa1602014. Epub 2016 Apr 4. PMID 27042964
- [Background] Chun KRJ, Brugada J, Elvan A, Geller L, Busch M, Barrera A, Schilling RJ, Reynolds MR, Hokanson RB, Holbrook R, Brown B, Schluter M, Kuck KH; FIRE AND ICE Investigators. The Impact of Cryoballoon Versus Radiofrequency Ablation for Paroxysmal Atrial Fibrillation on Healthcare Utilization and Costs: An Economic Analysis From the FIRE AND ICE Trial. J Am Heart Assoc. 2017 Jul 27;6(8):e006043. doi: 10.1161/JAHA.117.006043. PMID 28751544
- [Background] Andrade JG, Champagne J, Deyell MW, Essebag V, Lauck S, Morillo C, Sapp J, Skanes A, Theoret-Patrick P, Wells GA, Verma A; EARLY-AF Study Investigators. A randomized clinical trial of early invasive intervention for atrial fibrillation (EARLY-AF) - methods and rationale. Am Heart J. 2018 Dec;206:94-104. doi: 10.1016/j.ahj.2018.05.020. Epub 2018 Oct 18. PMID 30342299
- [Background] Kapa S, Epstein AE, Callans DJ, Garcia FC, Lin D, Bala R, Riley MP, Hutchinson MD, Gerstenfeld EP, Tzou W, Marchlinski FE, Frankel DS, Cooper JM, Supple G, Deo R, Verdino RJ, Patel VV, Dixit S. Assessing arrhythmia burden after catheter ablation of atrial fibrillation using an implantable loop recorder: the ABACUS study. J Cardiovasc Electrophysiol. 2013 Aug;24(8):875-81. doi: 10.1111/jce.12141. Epub 2013 Apr 11. PMID 23577826
- [Background] Manganiello S, Anselmino M, Amellone C, Pelissero E, Giuggia M, Trapani G, Giordano B, Senatore G, Gaita F. Symptomatic and asymptomatic long-term recurrences following transcatheter atrial fibrillation ablation. Pacing Clin Electrophysiol. 2014 Jun;37(6):697-702. doi: 10.1111/pace.12387. Epub 2014 Mar 25. PMID 24665920
- [Background] Reissmann B, Wissner E, Deiss S, Heeger C, Schlueter M, Wohlmuth P, Lemes C, Mathew S, Maurer T, Sohns C, Saguner A, Santoro F, Hayashi K, Riedl J, Ouyang F, Kuck KH, Metzner A. First insights into cryoballoon-based pulmonary vein isolation taking the individual time-to-isolation into account. Europace. 2017 Oct 1;19(10):1676-1680. doi: 10.1093/europace/euw233. PMID 28201538
- [Background] Kotecha D, Breithardt G, Camm AJ, Lip GYH, Schotten U, Ahlsson A, Arnar D, Atar D, Auricchio A, Bax J, Benussi S, Blomstrom-Lundqvist C, Borggrefe M, Boriani G, Brandes A, Calkins H, Casadei B, Castella M, Chua W, Crijns H, Dobrev D, Fabritz L, Feuring M, Freedman B, Gerth A, Goette A, Guasch E, Haase D, Hatem S, Haeusler KG, Heidbuchel H, Hendriks J, Hunter C, Kaab S, Kespohl S, Landmesser U, Lane DA, Lewalter T, Mont L, Nabauer M, Nielsen JC, Oeff M, Oldgren J, Oto A, Pison L, Potpara T, Ravens U, Richard-Lordereau I, Rienstra M, Savelieva I, Schnabel R, Sinner MF, Sommer P, Themistoclakis S, Van Gelder IC, Vardas PE, Verma A, Wakili R, Weber E, Werring D, Willems S, Ziegler A, Hindricks G, Kirchhof P. Integrating new approaches to atrial fibrillation management: the 6th AFNET/EHRA Consensus Conference. Europace. 2018 Mar 1;20(3):395-407. doi: 10.1093/europace/eux318. PMID 29300976
- [Background] Pokushalov E, Romanov A, Corbucci G, Artyomenko S, Turov A, Shirokova N, Karaskov A. Ablation of paroxysmal and persistent atrial fibrillation: 1-year follow-up through continuous subcutaneous monitoring. J Cardiovasc Electrophysiol. 2011 Apr;22(4):369-75. doi: 10.1111/j.1540-8167.2010.01923.x. Epub 2010 Oct 11. PMID 20958836